CLINICAL TRIAL: NCT02757534
Title: Domperidone for the Treatment of Chronic Nausea and Vomiting Secondary to Gastroparesis
Brief Title: Domperidone for Chronic Nausea and Vomiting
Status: No longer available | Type: Expanded Access
Sponsor: Yehudith Assouline-Dayan (Other)
Responsible Party: Sponsor-Investigator, Yehudith Assouline-Dayan, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201504713
Record Dates: First submitted 2015-06-09; First posted 2016-05-02 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Domperidone

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Domperidone — The study drug will be given to relieve the symptoms of gastroparesis, including nausea and vomiting.

SUMMARY:
The purpose of this study is to provide oral domperidone to patients with gastroparesis, between the ages of 18 and 60 years of age, who have failed standard treatment. Standard therapy at the University of Iowa is eating blended foods, liquid diet, Eryped syrup (125 mg TID) 30 minutes before meals, or reglan (20 mg BID).

DETAILED DESCRIPTION:
This is a compassionate use research study for a non-FDA approved drug. We are inviting patients to participate in this research study because they have nausea and vomiting related to gastroparesis and have failed standard therapy. The purpose of this research study is to prescribe patients with domperidone. Domperidone is considered investigational, which means that it has not been approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 18 - 60
3. Symptoms or manifestation secondary to gastroparesis such as vomiting, nausea, the feeling you are full after you start eating, bloating and abdominal pain.
4. Subjects must have a comprehensive evaluation to eliminate other causes of their symptoms which includes gastric emptying scintigraphy, esophagogastroduodenoscopy (EGD), and the patient's subjective symptoms.
5. Subject has signed informed consent for the administration of domperidone that informs the patient of potential adverse events including:

   * increased prolactin levels
   * extrapyramidal side effects
   * breast changes
   * cardiac arrhythmias including QT prolongation and death
6. Female subjects must be:

   * surgically sterile (have had a hysterectomy or bilateral oophorectomy, or tubal ligation)
   * if sexual active, practicing an effective method of birth control such as hormonal prescription oral contraceptives, progesterone implants or injections, contraceptive patch, intrauterine device, or maintenance of a monogamous relationship with a male partner who has been surgically sterilized by vasectomy. A double barrier method such as condoms, diaphragms, or cervical caps with spermicidal foam, cream, or gel may be used as a method of birth control

Exclusion Criteria:

1. History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation, atrial fibrilation and Torsade des Pointes, subjects with minor forms of ectopy (PACs) are not necessarily excluded
2. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged corrected QT interval (QTc) (QTc>450 milliseconds for males, QTc>470 milliseconds for females)
3. Clinically significant electrolyte disorders
4. Hepatic dysfunction
5. Renal insufficiency
6. Gastrointestinal hemorrhage or obstruction
7. Presence of a prolactinoma (prolactin-releasing pituitary tumor)
8. Pregnant or breast feeding female
9. Known allergy to domperidone

The following medications are prohibited during the study:

1. Antidepressants: doxepin (Adapin®, Sinequan®, Zonalon®), clomipramine (Anafranil®), amoxapine (Asendin®), trazodone (Desyrel®), venlafaxine (Effexor®), nefazodone (Serzone®), fluvoxamine (Luvox®), paroxetine (Paxil®), fluoxetine (Prozac®, Sarafem®), nefazodone (Serzone®), sertraline (Zoloft®), amitriptyline (Elavil®, Endep®, Etrafon®, Limbitrol®, Triavil®), maprotiline (Ludiomil®), desipramine (Norpramin®), nortriptyline (Pamelor®), trimipramine (Surmontil®), imipramine (Tofranil®), protriptyline (Vivactil®),
2. Anti-psychotics: haloperidol (Haldol®), chlorpromazine (Thorazine®, Ormazine®), chlorpromazine pimozide (Orap®), sertindole (Serlect®), quetiapine (Seroquel®), mesoridazine (Serentil®), perphenazine (Triavil®), fluphenazine (Apo-Fluphenazine®, Modecate Concentrate®, Moditen®, Permitil®, phenazine methosulfate-Fluphenazine®, Prolixin®, Rho-Fluphenazine®), promazine (Sparine®), trifluoperazine (Stelazine®)
3. Anti-Emetics: prochlorperazine (Compazine®), thioridazine (Mellaril®), promethazine (Phenergan®), mesoridazine (Serentil®), thiethylperazine, (Torecan®), perphenazine (Trilafon®), dolasetron (Anzemet®), dronabinol (Marinol®), droperidol (Inapsine®)
4. Anti-infective agents: erythromycin (such as E.E.S.®, E-Mycin®, Ilotycin® , Pediazole®, Akne-mycin®), clarithromycin (Biaxin®), troleandomycin (TAO®), norfloxacin (Ciproxin®, Noroxin®), quinine sulfate, quinupristin and dalfopristin (Synercid®), pentamidine (Nebupent®, Pentacarinat®, Pentam®), sparfloxacin (Zagam®), grepafloxacin (Raxar®), azithromycin (Zithromax®), ofloxacin (Floxin®). Levofloxacin (Levaquin®)
5. Anti-Fungal Agents: fluconazole (Diflucan®), itraconazole (Sporanox®), ketoconazole (Nizoral®), miconazole (Micatin®, Monistat®), terconazole (Terazol®), tioconazole (Vagistat®), butoconazole (Femstat 3®)
6. Antivirals: foscarnet (Foscavir®)
7. Protease Inhibitors: indinavir (Crixivan®), amprenavir (Agenerase®), ritonavir (Norvir®), nelfinavir (Viracept®), saquinavir (Invirase®, Fortovase®),
8. Anti-Hypertensives: nicardipine (Cardene®), isradipine (Dynacirc®), moexipril/ hydrochlorothiazide (HCTZ) (Uniretic®)
9. Calcium Channel Blockers: verapamil (Calan®), diltiazem (Cardizem®), diltiazem/enalapril (Teczem®), verapamil/trandolapril (Tarka®), tocainide (Tonocard®), bepridil (Vascor®)
10. Anti-Arrhythmics: disopyramide (Norpace®, Norpace Controlled Release ®), quinidine (such as Quinidex®, Cardioquin®, Quinaglute®, Duraquin®), procainamide (Procanbid® , Procan®, Pronestyl®,), flecainide (Tambocor®), sotalol (Betapace®), bretylium (Bretylol®), amiodarone (Cordarone®), ibutilide (Corvert®), moricizine (Ethmozine®)
11. Diuretics: bumetanide (Bumex®), furosemide (Lasix®), torsemide (Demadex®), ethacrynic Acid (Edecrin®), chlorothiazide (Diuril®), Indapamide (Lozol®)
12. Antilipemics: probucol (Lorelco®), Bepridil (Vascor®), mibefradil (Posicor®),
13. Hematological Agents: cilostazol (Pletal®)
14. Respiratory Agents: zafirlukast (Accolate®), salmeterol (Serevent®)
15. Gastrointestinal Agents: cimetidine (Tagamet®), cisapride (Propulsid®)
16. Antidiarrheal: octreotide (Sandostatin®)
17. Antihistamines: azelastine (Astelin®), clemastine (Tavist®)
18. Migraine treatment: naratriptan (Amerge®), sumatriptan (Imitrex®), zolmitriptan (Zomig®)
19. Antimalarial: halofantrine
20. Muscle relaxants: tizanidine (Zanaflex®)
21. Narcotic Dependence: levomethadyl (Orlaam®)
22. Miscellaneous: tamoxifen (Nolvadex®), warfarin (Coumadin®), phenytoin (Dilantin®), ziprasidone (Geodon®), risperidone (Risperdal®), formoterol fumarate (Foradil Aerolizer®), sildenafil (Viagra®)
23. Drugs that prolong the QT Interval: albuterol, alfuzosin, amantadine, amisulpride, amphetamine, arsenic trioxide, astemizole, atazanavir, atomoxetine, chloral hydrate, chloroquine, ciprofloxacin, citalopram, clozapine, cocaine, dexmethylphenidate, diphenhydramine, dobutamine, dofetilide, dopamine, dronedarone, ephedrine, epinephrine, eribulin, escitalopram, famotidine, felbamate, fenfluramine, fingolimod, fosphenytoin, galantamine, gatifloxacin, gemifloxacin, granisetron, iloperidone, isoproterenol, lapatinib, levalbuterol, lisdexamfetamine, lithium, metaproterenol, methadone, methylphenidate, midodrine, moxifloxacin, nilotinib, norepinephrine, ondansetron, oxytocin, paliperidone, perflutren lipid microspheres, phentermine, phenylephrine, phenylpropanolamine, protriptyline, pseudoephedrine, ranolazine, ritodrine, roxithromycin, sibutramine, solifenacin, sunitinib, tacrolimus, telithromycin, terbutaline, terfenadine, tolterodine, trimethoprim-sulfa, vandetanib, vardenafil, voriconazole.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yehudith Assouline-Dayan, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States